CLINICAL TRIAL: NCT04587375
Title: Diagnosis of Endocrine Dysfunctions in Covid-19 : Explorations of the Plasma Renin and Aldosterone Levels in Patients With Covid-19 Infection.
Brief Title: Diagnosis of Endocrine Dysfunctions in Covid-19
Acronym: Dyhor-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0205
Record Dates: First submitted 2020-06-18; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Covid 19
Keywords: Covid-19; Renin Angiotensin Aldosterone System; Hormon disorders
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As observed with SARS-CoV responsible for SARS 2003, the new coronarovirus SARS-CoV-2 uses the angiotensin converting enzyme type 2 (ACE2) as cellular receptor to infect cells. The renin aldosterone angiostensin system (RAAS) has known effects in the lungs: some receptors are pro-inflammatory, others are anti-inflammatory. Thus the deregulation of the RAAS induced by the SARS-CoV-2 could explain the inflammatory response of Covid-19 infection and be a modulator of the severity of its course.

Furthermore, the SARS 2003 experience suggests that there may be others endocrine involvment, particularly an failure on the hypothalamus-pituitary and adrenal axis. Indeeed, cases of hypocorticism and hypothyroidism of central origin were described.

Altogether, the endocrine system might play a role both in the pathophysiology of Covid-19 infection and in the activity and severity of the disease.

In this study, the investigators proposed to explore endocrine functions on biological samples in a series of patients admitted for Covid-19 in our clinic.

ELIGIBILITY:
Inclusion criteria:

- Patients with Covid-19 diagnosis and hospitalized in our clinic

Exclusion criteria:

- Minor patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Covid-19 diagnosis hospitalized in Montpellier University hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Plasma aldosterone levels | 1 day (at inclusion)
  Plasma aldosterone levels
Plasma renin levels | 1 day (at inclusion)
  Plasma renin levels

SECONDARY OUTCOMES:
covid-19 infection severity | 1 day (at inclusion)
  covid-19 infection severity : Ordinal scale of 7 values from 1 to 7 (1- not hospitalized, no limitation on activities; 2- not hospitalized, limitations on activities; 3- hospitalized, not requiring supplemental oxygen; 4- hospitalized, requiring supplemental oxygen; 5- hospitalized, on non-invasive ventilation or high flow oxygen devices; 6- hospitalized, on invasive mechanical ventilation or ECMO and 7- death).
Maximum severity of Covid-19 infection | 1 day (at inclusion)
  Maximum severity of Covid-19 infection using a seven-category ordinal scale at at the end of hospitalization : Ordinal scale of 7 values from 1 to 7 (1- not hospitalized, no limitation on activities; 2- not hospitalized, limitations on activities; 3- hospitalized, not requiring supplemental oxygen; 4- hospitalized, requiring supplemental oxygen; 5- hospitalized, on non-invasive ventilation or high flow oxygen devices; 6- hospitalized, on invasive mechanical ventilation or ECMO and 7- death).
Plasma aldosterone level | 1 day (at the end of hospitalization)
  Plasma aldosterone level
Plasma ACTH level | 1 day (at the end of hospitalization)
  Plasma ACTH level
Plasma cortisol level | 1 day (at inclusion)
  Plasma cortisol level
Plasma cortisol level | 1 day (at the end of hospitalization)
  Plasma cortisol level
Plasma T3l level | 1 day (at the end of hospitalization)
  Plasma T3l level
Plasma T3l level | 1 day (at inclusion)
  Plasma T3l level
Plasma ACTH level | 1 day (at inclusion)
  Plasma ACTH level
Plasma LH level | 1 day (at inclusion)
  Plasma LH level
Plasma LH level | 1 day (at the end of hospitalization)
  Plasma LH level
Plasma DHEA level | 1 day (at the end of hospitalization)
  Plasma DHEA level
Plasma DHEA level | 1 day (at inclusion)
  Plasma DHEA level
Plasma estradiol (female) or testosterone (male) level | 1 day (at the end of hospitalization)
  Plasma estradiol (female) or testosterone (male) level
Plasma estradiol (female) or testosterone (male) level | 1 day (at inclusion)
  Plasma estradiol (female) or testosterone (male) level
Plasma FSH level | 1 day (at the end of hospitalization)
  Plasma FSH level
Plasma FSH level | 1 day (at inclusion)
  Plasma FSH level
type of treatments | 1 day
  type of treatments
Clinical characteristics | 1 day
  Clinical characteristics extracted from electronic medical
radiological characteristics | 1 day
  radiological characteristics : quantification of the percentage of lesional damage to the pulmonary parenchyma

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GUILPAIN, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC